CLINICAL TRIAL: NCT02513368
Title: Peri Implant Soft Tissue Healing in Single Implant Restoration Using the Guided Bone Regeneration Technique Ore a Connective Tissue Graft
Brief Title: Peri Implant Soft Tissue Healing in Single Implant Restoration Using Two Different Techniques
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Firenze and Siena, Napoli, Italy (Other)
Responsible Party: Principal Investigator, nicola baldini, oral surgeon, University of Firenze and Siena, Napoli, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHSIR
Record Dates: First submitted 2015-07-03; First posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Oral Soft Tissue Conditions
Keywords: aesthetic; connective tissue graft; mucosa thickness

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bio-Oss®, Bio-Gide® (Experimental): augmentation procedure with Bio-Oss® and Bio-Gide®
  Interventions: Device: augmentation procedure with Bio-Oss® and Bio-Gide®
- connective tissue graft (Active Comparator): augmentation procedure with connective tissue graft
  Interventions: Procedure: augmentation procedure with connective tissue graft

INTERVENTIONS:
Device: augmentation procedure with Bio-Oss® and Bio-Gide® — soft tissue management using GBR procedure
  Arms: Bio-Oss®, Bio-Gide®
Procedure: augmentation procedure with connective tissue graft — soft tissue management using the bilaminar technique
  Arms: connective tissue graft

SUMMARY:
The aim of the present study was to propose the employment of Bio-Oss® and Bio-Gide® at implant site in order to evaluate if the increased bucco-lingual bone thickness could enhance the stability of peri implant soft tissue, when compared to the grafting technique ( bilaminar technique), performed in association with implant placement .

DETAILED DESCRIPTION:
With respect to the soft tissue management many surgical approaches have been described in order to increase soft tissue volume and keratinized tissue height at implant site: roll flaps, connective tissue graft , epithelial connective tissue graft. In recent years, soft tissue substitutes , such as acellular dermal matrix or collagen matrix have been proposed to increase the dimensions of peri implant soft tissues; however, further studies have demonstrated that the allograft materials were less effective and less predictable than autogenous soft tissue grafts, in terms of increasing attached keratinized tissue , due to the considerable shrinkage and inconsistent quality of the attached tissue gained ; consequently soft tissue graft from the palate are currently considered the gold standard for augmenting peri implant soft. Some clinical studies proposed the association of contour augmentation by guided bone regeneration (GBR) with implant placement. The aim of these procedures is to restore the missing volume and to establish a facial bone wall of sufficient height and thickness to serve as a support for peri implant soft tissues; in these terms, GBR could be considered important to increase the stability of peri implant soft tissue , preventing the marginal soft tissue shrinkage and the following exposition of implant . This could be a valid approach to stabilize coronal peri implant soft tissue and at the same time less traumatic than grafting procedures.

ELIGIBILITY:
Inclusion Criteria:

* one missing tooth in the anterior maxilla
* facial keratinized mucosa thickness of at least 2mm

Exclusion Criteria:

* heavy smokers
* systemic diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
change from baseline in the clinical characteristics of the peri implant mucosa | one month and one year after the placement of the definitive crowns
  Buccal mucosa thickness was assessed with a calibrated endodontic file, 2 mm apical to the bone crest

SECONDARY OUTCOMES:
Change from baseline in probing pocket depth recorded at both mesial and distal tooth , adjacent to the implant site, by means of a periodontal probe | one month and one year after the placement of the definitive crowns
change from baseline in height of keratinised tissue recorded at both mesial and distal tooth , adjacent to the implant site , by means of a periodontal probe | one month and one year after the placement of the definitive crowns

CONTACTS AND LOCATIONS:
Overall Officials: massimo de sanctis, dentist, Principal Investigator — school of dentale medicine , university of siena
Locations (2):
- Italy (2):
  - Siena University, Department of Periodontology, Policlinico Le Scotte Siena., Siena, Siena
  - Tuscan School of Dentistry, Siena, Siena

REFERENCES:
- [Background] Buser D, Chappuis V, Bornstein MM, Wittneben JG, Frei M, Belser UC. Long-term stability of contour augmentation with early implant placement following single tooth extraction in the esthetic zone: a prospective, cross-sectional study in 41 patients with a 5- to 9-year follow-up. J Periodontol. 2013 Nov;84(11):1517-27. doi: 10.1902/jop.2013.120635. Epub 2013 Jan 24. PMID 23347346